CLINICAL TRIAL: NCT00817297
Title: Cross-over Comparison of the V60 System to Other Bi-Level Noninvasive Ventilators for Adult Patients With Respiratory Failure or Respiratory Insufficiency
Brief Title: Cross-over Comparison of the V60 System to Other Bi-Level Noninvasive Ventilators
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Respironics, California, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: V60-1050767VP v 2.4
Record Dates: First submitted 2009-01-03; First posted 2009-01-06 (Estimated); Last update posted 2017-11-17 (Actual); Status verified 2017-04

CONDITIONS: Respiratory Insufficiency; Respiratory Failure
Keywords: noninvasive ventilation
MeSH Terms: conditions — Respiratory Insufficiency

STUDY DESIGN:
Who Masked: Participant
Masking Description: Subject was blinded to device identity
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- V60 Mask, Then Conventional Mask (Other): Experimental V60 Mask Ventilator for treating adult patients with COPD, then Comparator Conventional Mask Ventilator for treating adult patients with COPD
  Interventions: Device: noninvasive ventilator
- Conventional Mask, Then V60 Mask (Other): Comparator Conventional Mask noninvasive Ventilator for treating adult patients with COPD, then Experimental V60 Mask noninvasive Ventilator for treating adult patients with COPD.
  Interventions: Device: noninvasive ventilator

INTERVENTIONS:
Device: noninvasive ventilator — Experimental V60 Mask noninvasive Ventilator for treating patients with COPD, then Comparator Conventional Mask noninvasive Ventilator for treating patients with COPD in crossover study design

SUMMARY:
The purpose of this study is to compare a new noninvasive ventilator to existing ventilators already used for patient care.

DETAILED DESCRIPTION:
The primary objective of this study was to compare the performance (i.e., patient self-reported Comfort score) of the V60 device and a conventional noninvasive ventilator (patient's current ventilator). For the User Needs Assessment, the primary objective of the study was to validate the V60 to user needs. All patients were volunteers from the Respiratory Section of the Health Sciences Centre at the University of Manitoba. The study utilized a randomized 2-period cross-over study design to compare the V60 System to the patients' existing conventional noninvasive ventilator in different ventilation modes.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years and < 85 years
* Weight > 20 kg (44 lbs)
* Respiratory failure or respiratory insufficiency
* Ability to cooperate with the investigators

Exclusion Criteria:

* An endotracheal tube or tracheostomy in place
* Hemodynamic instability
* Prolonged apnea
* Inability to maintain the airway
* A recent history of cardiac and or respiratory arrest
* Acute hemorrhage
* Multiple organ system failure
* Undrained pneumothorax
* High risk for aspiration
* Metastatic or terminal cancer
* Do-not-resuscitate orders
* Inability to clear respiratory secretions
* Inability to fit a mask
* Facial surgery, trauma, or deformity
* Upper gastrointestinal or airway surgery
* Pregnancy
* Refractory delirium
* Inability or unwillingness to provide Informed Consent
* PaO2 < 50 mmHg

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2009-01-17 (Actual); Primary Completion 2009-03-03 (Actual); Study Completion 2009-04-07 (Actual)

PRIMARY OUTCOMES:
Breathing comfort | 0, 15, and 30 minutes

SECONDARY OUTCOMES:
Physiological variables | 0, 15, and 30 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Steven Mink, MD, Principal Investigator — University of Manitoba, Winnipeg, Manitoba, Canada
Locations (1):
- GF-221 Health Sciences Centre, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No